CLINICAL TRIAL: NCT02158624
Title: The Correlation for Improvement of Visual Acuity and QOL After Ranibizmab Treatment for Age-Related Macular Degeneration Patients
Brief Title: Ranibizumab Treatment for Age-Related Macular Degeneretion
Acronym: QUATRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyushu University (Other)
Collaborators: University of Occupational and Environmental Health (Other); Kurume University (Other); Fukuoka University (Other); Clinical Research Support Center Kyush (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Yuji Oshima, Assistant professor, Kyushu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-E-09
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Visual Disorder Due to Age-related Macula Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: Intravitreal Lucentis 0.5mg

INTERVENTIONS:
Drug: Intravitreal Lucentis 0.5mg

SUMMARY:
To establish the correlation between visual acuity improvement and QOL measurement after ranibizumab treatment for AMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Active primary or recurrent subfoveal choroidal neovascularization lesion due to AMD
* Subjects of either gender age 50 years or older
* Visual acuity better than 0.05 decimal( 20/400 Snellen)
* Signed informed consent form

Exclusion Criteria:

* Prior treatment for neovascular AMD in the study eye, for example, PDT or anti-VEGF therapy
* Patients whose lesion site evaluated by FA examination is more than 12DA in subject eye
* Patients with treatment of triamcinolone intravitreal injection within 6 months in subject eye
* Patients with a history of intraocular surgical operation(including cataract)within 3 months in subject eye
* Patients with serious allergic history to such as fluorescein, indocyanine green, iodophors
* The pregnant or lactating woman

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Baseline change of visual acuity and QOL after ranibizumab treatment | 3 months
  Analyze the correlation between visual acuity improvement and QOL assessment using VFQ-25 and Patient Satisfaction Questionnaire before and after initial ranibizumab treatment for AMD patients.

SECONDARY OUTCOMES:
To evaluate the correlation between the changes of visual acuity and QOL measurement during one year follow-up observations | 1year

OTHER OUTCOMES:
Baseline change of central retinal thickness by OCT examination. | 3 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Kyushu University Hospital, Maidashi, Higashiku, Fukuoka-city, Fukuoka, Japan